CLINICAL TRIAL: NCT01421784
Title: Investigating the Feasibility of Using Rapid Cine-MRI for Monitoring Moving and Deforming Tumors
Brief Title: Using Rapid Cine-MRI for Monitoring Moving and Deforming Tumors
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left the institution
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STU 042011-034
Record Dates: First submitted 2011-08-10; First posted 2011-08-23 (Estimated); Last update posted 2020-08-20 (Actual); Status verified 2018-06

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cine-MRI (Other): Rapid Cine-MRI
  Interventions: Other: cine MRI

INTERVENTIONS:
Other: cine MRI — Rapid Cine-MRI for Monitoring Moving and Deforming Tumors

SUMMARY:
In this study, the researchers investigate the feasibility of using rapid cine MR imaging to provide both offline and online soft-tissue-based image guidance. Such images will provide a significantly more complete picture of the spatial and temporal changes in thoracic anatomy. This more complete information will lay the groundwork for better radiotherapy planning and dose delivery in the presence of respiratory motion.

DETAILED DESCRIPTION:
Rapid MRI scans from Stage I-IV non-small-cell lung cancer (NSCLC) patients will be acquired. MR acquisition will be performed without extrinsically administered contrast, using a balanced turbo field echo (TFE) sequence and commercially available coils.

ELIGIBILITY:
Inclusion Criteria:

* AJCC Stage I, II, III or IV non-small-cell lung cancer to be treated using radiotherapy will be eligible for this study.
* Any types and amounts of prior therapy will be allowed for this study.
* Subjects must be greater than or equal to 18 years of age. There are no gender or ethnic restrictions.
* Ability to understand and the willingness to sign a written informed consent document.
* Able to tolerate supine position
* ECOG performance status of 3 or less

Exclusion Criteria:

* MRI-incompatible metallic implants, embedded metallic objects, implanted biomedical devices e.g., cardiac pacemakers
* Women who are pregnant or trying to get pregnant
* Pain in supine position

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2011-09 (Actual); Primary Completion 2015-11-25 (Actual); Study Completion 2015-11-25 (Actual)

PRIMARY OUTCOMES:
To measure time series of MRI imaging by the b-SSFP sequence. | 6 weeks
  To use fast acquisition sequences to obtain 2D and 3D cine MR images of moving and deforming lung tumors. The signal to noise ration (SNR) and spatiotemporal resolution of imaging sequences will be optimized into a format potentially useful for radiotherapy guidance.

CONTACTS AND LOCATIONS:
Overall Officials: Amit Sawant, Ph.D., Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States